CLINICAL TRIAL: NCT05577845
Title: Safety & Efficacy of 5-HT3 Receptor Antagonist (Ramosetron) Versus Loperamide for the Treatment of Low Anterior Resection Syndrome (RALLARS): Multicenter Randomized Controlled Trial
Brief Title: 5-HT3 Receptor Antagonist (Ramosetron) vs Loperamide for the Treatment of Low Anterior Resection Syndrome(RALARS)
Acronym: RaLARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ryoo, Seung-Bum, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2208-086-1351
Record Dates: First submitted 2022-09-28; First posted 2022-10-13 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: LARS - Low Anterior Resection Syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ramosetron (Experimental)
  Interventions: Drug: Ramosetron
- Loperamide (Active Comparator)
  Interventions: Drug: Ramosetron

INTERVENTIONS:
Drug: Ramosetron — Ramosetron, 4 weeks

SUMMARY:
Safety & Efficacy of 5-HT3 Receptor Antagonist (Ramosetron) versus Loperamide for the Treatment of Low Anterior Resection Syndrome (RALLARS): Multicenter Randomized Controlled Trial

ELIGIBILITY:
Inclusion Criteria:

* mid and low rectal cancer (AV<15cm)
* stage II, III, preop long-course CCRT, then ileostomy repair
* about 1~12 months after operation (no stomy)
* about 1~6 months after ileostomy repair
* major LARS

Exclusion Criteria:

* recurred rectal cancer
* stage IV
* IBD
* uncontrolled preoperative fecal incontinence or constipation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 212 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
major Low Anterior Resection Syndrome (LARS) | 0 weeks
  LARS score (0-20, no, 21-29, minor, 30-42, major)
Difference of improvement of major Low Anterior Resection Syndrome (LARS) | 4 weeks
  LARS score (0-20, no, 21-29, minor, 30-42, major)

SECONDARY OUTCOMES:
EORTC QLQ-C30 score | 0 weeks
  Quality of life surveillance
EORTC QLQ-C30 score | 4 weeks
  Quality of life surveillance

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongro-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided